CLINICAL TRIAL: NCT07329647
Title: The Neurovascular Coupling as a Target for Cognitive Enhancement in Vascular Cognitive Decline Through an Innovative Nitrate-driven Dietary Supplementation.
Brief Title: Targeting Neurovascular Coupling in Cognitive Decline Via Nitrate-Based Supplementation
Acronym: DietNOBrain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Coimbra (Other)
Responsible Party: Principal Investigator, Miguel Castelo-Branco, Professor, University of Coimbra
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: DietNOBrain01CNC; 2022.05454.PTDC (Other Grant/Funding Number: Fundação para a Ciência e Tecnologia (FCT))
Record Dates: First submitted 2025-11-17; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-11

CONDITIONS: Small Vessel Cerebrovascular Disease; Diabete Mellitus
MeSH Terms: conditions — Cerebral Small Vessel Diseases; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nitrate rich beetroot juice (Experimental)
  Interventions: Dietary Supplement: Beetroot Juice - Active
- Nitrate depleted beetroot juice (Placebo Comparator)
  Interventions: Dietary Supplement: Beetroot Juice - Placebo

INTERVENTIONS:
Dietary Supplement: Beetroot Juice - Active — 140 ml beetroot juice/day, corresponding to approximately 0.8 g of nitrate that will constitute a period of 2 weeks with a nitrate-diet (beetroot).
  Arms: Nitrate rich beetroot juice
Dietary Supplement: Beetroot Juice - Placebo — 140 ml nitrate-depleted beetroot juice/day, that will constitute a period of 2 weeks with a nitrate-depleted diet (beetroot).
  Arms: Nitrate depleted beetroot juice

SUMMARY:
Diet is established among the most relevant adjustable variables of human health in modern societies. The recognition by the World Health Organization of cognitive impairment and dementia associated with aging as one of the major public health challenges of our time, highlights the imperative need for a more comprehensive understanding of how different aspects of lifestyle, in particular diet, affect neural function and consequent cognitive performance throughout lifespan.

The brain is endowed with fine mechanisms for a precise spatial and temporal control of cerebral blood flow (CBF) according to neural activity, the neurovascular coupling (NVC). Mounting evidence from preclinical and human studies demonstrate that NVC dysfunction is a key early factor contributing to the pathogenesis of cognitive decline and vascular cognitive impairment (VCI) in aging and conditions associated with accelerated microvascular aging, such as cerebral small vessel disease (cSVD). Failure at any part of the NVC pathway disrupts CBF resulting in catastrophic depletion of oxygenation and energy supply to brain cells, and, in the long run, to neuronal dysfunction and cognitive impairment.

The investigators have shown that nitric oxide (NO) synthesized by neuronal nitric oxide synthase (nNOS) is a direct mediator of NVC and that decreased bioavailability of NO along aging compromised NVC and reduced local CBF. Shortly after the identification of nNOS as a source of NO for vasodilation in the brain, an alternative pathway for NO production independent of nNOS, relying on the sequential reduction of nitrate, the nitrate:nitrite:NO pathway, was unveiled.

Nitrate consumed in green leafy vegetables as part of a normal diet is bioactivated to nitrite and both compounds are permanent constituents of blood/tissues in animal species, influencing CBF and resulting in improvements in learning and memory in rodents and VCI patients. However, a critical question remains on whether NO produced from nitrite is functionally linked to neuronal activation. This is key to understanding whether dietary nitrate can be linked to neuronal-dependent CBF increases and cognitive performance.

The investigators and others have shown that upon excitatory stimulation, ascorbate is released from neurons being available for nitrite reduction and our preliminary data supports that NO bioavailability and CBF might be maintained independently of nNOS by the reduction of nitrite to NO in the brain extracellular space upon neuronal activation (unpublish data). This innovative mechanism functionally links the production of NO from nitrite to neuronal activation, triggering CBF increases and maintaining an operative NVC. A further facet is that, bridging diet and cognitive performance, this mechanism incorporates modulatory elements which is open to adjustment by diet via nitrate.

Thus, in this pilot trial a proof of concept study will be conducted to investigate the clinical impact of a dietary nitrate supplementation intervention in a clinical population with VCI due to small vessel disease, as measured by changes on NVC and cognitive performance.

The investigators hypothesise that functional NVC is maintained operative in VCI patients by increasing NO bioavailability in the extracellular space of the brain through a nitrate -rich diet that, in turn, supports an adequate CBF in response to neuronal activation, modulating the molecular mechanisms and cognitive performance of disease-related physiological and cognitive markers.

DETAILED DESCRIPTION:
Professor João Laranjinha (CNC-UC) is the lead scientific contributor of the study.

ELIGIBILITY:
Inclusion Criteria:

* Formal diagnosis of cerebral small vessel disease (grades 1 to 3 in the Age-Related White Matter Changes Scale as assessed by Computerized Tomography or Magnetic Ressonance Imaging - MRI) and patients at high risk for cerebral small vessel disease with diabetes mellitus;
* Subject has capacity and is capable of giving written informed consent;
* Subject is able to read, comprehend and record information written in Portuguese.

Exclusion Criteria:

* Vascular diseases other than cerebral Small Vessel Disease (cSVD);
* Stroke event less than 6 months ago;
* Unsuitable for MRI scanning because of presence of any standard MRI contraindication (e.g presence of a cardiac pacemaker, other medical implants or devices, or the presence of ferromagnetic metal foreign bodies);
* Needle phobia;
* Inability or intolerance to dietary polyphenol adjustment;
* Current smoker;
* Alcohol abuse, drug abuse or use of drugs affecting cognitive assessment, such as sedatives, hypnotics, nootropic drugs, cholinergic drugs;
* Use of medications that may be contraindicated or interact with the high nitrate diet, such as nitroglycerin or nitrate preparations used for angina, or phosphodiesterase type 5 (PDE5) inhibitors, including sildenafil (Viagral);
* Patients previously diagnosed with dementia;
* Presence of congenital mental retardation and severe neurological and psychiatric diseases;
* Illiterate or severe visual or hearing impairment that may prevent patients from cooperating with cognitive assessment;
* Relevant depression or other unrelated serious mental illness;
* Severe cardiac, pulmonary, renal or hepatic insufficiency;
* Patients who have participated in other interventional clinical studies within the last 3 months, or are participating in other interventional clinical studies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-05-09 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Memory retrieval cognitive task (d prime) | From baseline to the end of treatment up to Week 4 and from baseline to the end of placebo up to Week 11.
  Comparing changes from baseline after dietary nitrate supplementation (standardised beetroot juice) during 14 days versus the placebo condition.
Memory encoding Blood Oxigenation Level Dependent (BOLD) signal amplitude | From baseline to the end of treatment up to Week 4 and from baseline to the end of placebo up to Week 11.
  Comparing changes from baseline after dietary nitrate supplementation (standardised beetroot juice) during 14 days versus the placebo condition.

SECONDARY OUTCOMES:
Ascorbate concentration in the posterior cingulate cortex | From baseline to the end of treatment up to Week 4 and from baseline to the end of placebo up to Week 11.
  Comparing changes in ascorbate concentration from baseline to after dietary nitrate supplementation (standardised beetroot juice) during 14 days versus the placebo condition.
Score on the Visual Analogue Scale of the health-related quality of life EQ-5D-5L questionnaire | From baseline to the end of treatment up to Week 4 and from baseline to the end of placebo up to Week 11.
  Comparing changes from baseline after dietary nitrate supplementation (standardised beetroot juice) during 14 days versus the placebo condition on the score of the Visual Analogue Scale of EQ-5D-5L questionnaire, ranging from 0 to 100, where higher values mean better health related quality of life.
Nitrate concentration in the blood | From baseline to the end of treatment up to Week 4 and from Week 7 to the end of placebo up to Week 11.
  Comparing changes in nitrate concentration from baseline to after dietary nitrate supplementation (standardised beetroot juice) during 14 days versus the placebo condition.
Glutathione concentration in the posterior cingulate cortex | From baseline to the end of treatment up to Week 4 and from baseline to the end of placebo up to Week 11.
  Comparing changes in glutathione concentration from baseline to after dietary nitrate supplementation (standardised beetroot juice) during 14 days versus the placebo condition.
N-acetylaspartate concentration in the posterior cingulate cortex | From baseline to the end of treatment up to Week 4 and from baseline to the end of placebo up to Week 11.
  Comparing changes in n-acetylaspartate concentration from baseline to after dietary nitrate supplementation (standardised beetroot juice) during 14 days versus the placebo condition.
Glutamate concentration in the posterior cingulate cortex | From baseline to the end of treatment up to Week 4 and from baseline to the end of placebo up to Week 11.
  Comparing changes in glutamate concentration from baseline to after dietary nitrate supplementation (standardised beetroot juice) during 14 days versus the placebo condition.
Gamma-aminobutyric acid (GABA) concentration in the posterior cingulate cortex | From baseline to the end of treatment up to Week 4 and from baseline to the end of placebo up to Week 11.
  Comparing changes in gamma-aminobutyric acid (GABA) concentration from baseline to after dietary nitrate supplementation (standardised beetroot juice) during 14 days versus the placebo condition.
Lactate concentration in the posterior cingulate cortex | From baseline to the end of treatment up to Week 4 and from baseline to the end of placebo up to Week 11.
  Comparing changes in lactate concentration from baseline to after dietary nitrate supplementation (standardised beetroot juice) during 14 days versus the placebo condition.
Creatine concentration in the posterior cingulate cortex | From baseline to the end of treatment up to Week 4 and from baseline to the end of placebo up to Week 11.
  Comparing changes in creatine concentration from baseline to after dietary nitrate supplementation (standardised beetroot juice) during 14 days versus the placebo condition.
Nitrite concentration in the blood | From baseline to the end of treatment up to Week 4 and from Week 7 to the end of placebo up to Week 11.
  Comparing changes in nitrite concentration from baseline to after dietary nitrate supplementation (standardised beetroot juice) during 14 days versus the placebo condition.
S-nitrosothiols concentration in the blood | From baseline to the end of treatment up to Week 4 and from Week 7 to the end of placebo up to Week 11.
  Comparing changes in S-nitrosothiols concentration from baseline to after dietary nitrate supplementation (standardised beetroot juice) during 14 days versus the placebo condition.

CONTACTS AND LOCATIONS:
Locations (2):
- Portugal (2):
  - Institute for Nuclear Sciences Applied to Health (ICNAS), University of Coimbra, Coimbra
  - Unidade de Saúde Local de Coimbra (ULS Coimbra), Coimbra

IPD SHARING:
Plan to Share IPD: Undecided